CLINICAL TRIAL: NCT02282644
Title: Individual Phenotype Analysis in Patients With Castration-Resistant Prostate Cancer With CellSearch® and Flow Cytometry
Acronym: PROMET II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013.824
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CellSearch (Experimental)
  Interventions: Biological: Bone marrow sampling

INTERVENTIONS:
Biological: Bone marrow sampling

SUMMARY:
The recent data suggest that cancer cells at the origin of prostate cancer metastases can be detected in an early stage. Available techniques allow phenotypic analysis of cancer cells in circulating blood (cellsearch) or in marrow hematopoietic (flow cytometry). Pilot study on 180 patients infected by prostate cancer at all stage of disease, show that c-met marker , integrin alpha 2 and 6 expressed in marrow and quantified by flow cytometry were predictor of metastatic progress. In this new study the investigators will analyze antibody panel by cellsearch and flow cytometry on marrow sample of castration-Resistant prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma or prostate
* Ongoing effective androgen deprivation therapy (testosterone ≤ 50 ng/mL)
* Castration-Resistant prostate cancer patient : defined as a minimum of 3 rising PSA values assessed and/or radiological progress confirmed by RECIST and PCWG2
* Patient who signed informed consent

Exclusion Criteria:

* Severe disorders of coagulation
* Major skin lesion on iliac crests
* Allergies in local anesthetics
* Psychological instability or psychiatric histories
* Uncertain follow-up and distant residence
* History of another invasive cancer and hematologic disease
* Patient deprived of their freedom by court or administrative order
* Revocation of consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Risk of death according to positive makers | Two years

SECONDARY OUTCOMES:
Risk of clinical progression according to positive markers. | Two years
Risk of biological progression according to positive markers. | Two years
Risk of radiological progression according to positive markers. | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot - service d'urologie, Lyon, France